CLINICAL TRIAL: NCT05534906
Title: The Detection of Small Early Liver Cancer With Natural History Follow up
Acronym: SELINA
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Cancer Research UK (Other); Roche Diagnostic Ltd. (Industry); OncImmune Ltd (Unknown); Perspectum (Industry); University of Nottingham (Other); Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Other Study IDs: SELINA
Record Dates: First submitted 2022-08-01; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Blood Specimen Collection; X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Small HCC with Cirrhosis: 200 patients diagnosed with small HCC (as defined in Eligibility Criteria) and cirrhosis
  Interventions: Other: Blood & Urine Samples
- Small HCC without Cirrhosis: 50 patients diagnosed with small HCC (as defined in Eligibility Criteria) but without cirrhosis
  Interventions: Other: Blood & Urine Samples
- Imaging Subgroup: In a subgroup of patients (N=80, around 64 patients with HCC with liver cirrhosis and around 16 patients with HCC without liver cirrhosis), additional magnetic resonance liver imaging & elastography will be performed
  Interventions: Other: Imaging

INTERVENTIONS:
Other: Blood & Urine Samples — Blood and urine samples will be collected to help identify biomarkers that can be used to detect liver cancer at the earliest possible time
  Groups: Small HCC with Cirrhosis; Small HCC without Cirrhosis
Other: Imaging — MRI & MRE Scans
  Groups: Imaging Subgroup

SUMMARY:
The SELINA study will recruit 200 patients with cirrhosis and small HCC and 50 patients with HCC but without cirrhosis (most of whom are expected to have FLD). Blood, urine and liver tissue samples (where available) will be collected for laboratory analysis. In a subgroup of patients (N=80, around 64 patients with HCC with liver cirrhosis and around 16 patients with HCC without liver cirrhosis), additional magnetic resonance liver imaging will be performed. The findings of the SELINA study aim to identify biomarkers that can be used to detect liver cancer at the earliest possible time, something we expect will increase the survival rate of HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study.
2. Male or Female aged 18 years or above.
3. Diagnosed with small HCC (Barcelona Clinic Liver Cancer Staging Criteria (BCLC) stage 0/A; 1-3 nodules <3cm, preserved liver function, performance status 0) with liver cirrhosis from any aetiology
4. Diagnosed with small HCC (as above) and without cirrhosis
5. Diagnosis of small HCC shown or confirmed within 3 months of study Visit 1
6. Patients with a diagnosis of HCC that was fully ablated or resected more than 6 months ago and now presenting with a new diagnosis of HCC in a different site in the liver may be included in the study
7. Histological confirmation is required to establish the diagnosis of HCC in patients without cirrhosis (imaging alone is not considered sufficient to establish the diagnosis of HCC).

Exclusion Criteria:

1. Patients judged by the investigator to be unsuitable for inclusion in the study (e.g. where the investigator feels that the participant will not be able to comply with the study procedures)
2. HCC with liver cirrhosis at BCLC stage B/C
3. Patients who have had a previous liver transplant (note, it is permitted to enrol patients on the liver transplant waiting list if they fulfil all inclusion/exclusion criteria)
4. Participants of the Pearl study
5. Patients who have had a previous diagnosis of HCC followed by therapy, and now have a recurrence at the same site in the liver
6. Patients who have received HCC specific therapy 3 months prior to study visit 1 (including resection, ablation [microwave/radiofrequency]), transarterial chemoembolization [TACE], select internal radiation therapy [SIRT] or stereotactic body radiation therapy [SBRT] 3, chemotherapy, immune modulators and other experimental therapies).

Exclusion Criteria for Imaging Subgroup

1. Any contra-indication to Magnetic Resonance Imaging (MRI) (e.g. claustrophobia, metal implants/fragments, implants, pregnancy, other conditions the scanner operator deems unsafe for MR scanning).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with small HCC with cirrhosis (N=200) or with HCC but without cirrhosis (N=50) aged 18 years and above
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2035-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Biomarkers associated with small HCC (Early detection [EDx] biomarkers) | Throughout study to completion; up to 5 years
  Classification performance metrics of EDx biomarkers, in cirrhosis patients with small HCC compared to non-HCC cirrhosis patients

SECONDARY OUTCOMES:
Prognostic ability of Early Detection (EDx) bio-markers | Throughout study to completion; up to 5 years
  Ability of EDx biomarkers to discriminate between individuals who go onto develop adverse outcomes (e.g. HCC rapid tumour progression, liver decompensation, liver related mortality, liver transplantation) versus those who do not. Measured via Harrell's concordance index and Royston's D statistic.
Whether combinations of EDx tests improve the diagnostic and prognostic performance | Throughout study to completion; up to 5 years
  Model fit statistics comparing univariate and multivariate models, including Harrell's adequacy index. The change in model discrimination (e.g. Delta Concordance-index and Delta D-statistic) will also be considered.
Proportion of patients with HCC events according to time since treatment with curative intent. | Throughout study to completion; up to 5 years
  To study the natural history of small HCC. Proportion of patients with HCC recurrence, all-cause mortality, liver mortality etc, according to time since treatment with curative intent..

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Barnes, Principal Investigator — University of Oxford
Locations (1):
- Hepatology Clinical Trial Unit, John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- See also: DeLIVER Project Website — https://deliver.cancer.ox.ac.uk/